CLINICAL TRIAL: NCT04079153
Title: Effects of Two Different Amounts of Mandibular Protrusion in Obstructive Sleep Apnea Patients Using Mandibular Advancement Appliance : A Randomized Controlled Trial
Brief Title: Effects of Two Different Amounts of Mandibular Protrusion in OSA Patients Using Mandibular Advancement Appliance
Acronym: MAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Chin Mei H'uah, Postgraduate Student, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019421-7342
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: mandibular advancement appliance, protrusion
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Group A will be assigned for intervention group, whereby patients will receive their MAA set at 25% of mandibular maximal protrusion while Group B will be assigned for control group, whereby patients will receive their MAA set at 50% of mandibular maximal protrusion.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to the intervention allocation and intervention group. A single orthodontic resident will treat all the patients, and one dental technician will construct all the appliances. The clinician, however, is unable to be blinded due to the need to prescribe the MAA as being randomized. Data collection and analysis will be done by the orthodontic resident. Blinding during data collection will not possible but after data collection, all the data will be coded before being processed and analysed, ensuring blinding of this stage of study. Sleep technician and physician who respectively carried out and analysed the polysomnography will be blinded to the treatment assignment. Statistician who analysed the data will also blinded to the group of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25% of maximal mandibular advancement (Active Comparator): 25% of maximal mandibular advancement of individual protrusion range
  Interventions: Device: Mandibular advancement Appliance
- 50% of maximal mandibular advancement (Active Comparator): 50% of maximal mandibular advancement of individual protrusion range
  Interventions: Device: Mandibular advancement Appliance

INTERVENTIONS:
Device: Mandibular advancement Appliance — Advances the mandible at desired range at a fixed vertical dimension

SUMMARY:
Obstructive sleep apnea (OSA) is a complex disease associated with repeated closure of the upper airway during sleep which causes excessive daytime sleepiness. Daytime sleepiness can affects daytime performance undesirably and reduces driving performance causing an increased risk for accidents. It can also lead to high blood pressure, strokes, and eventually death.

Until now, there is no standardize value for the jaw advancement for the mandibular advancement appliance. It was found that when comparing the jaw advancement amount of 50% and above 50%, there is no additional efficacy. Efficacy of jaw advancement below 50% is lacking. Patients usually experience more complications with more advancement, there the investigators need to study the optimal mandibular advancement with least complication to the patients.

DETAILED DESCRIPTION:
This is a single-center, double blind (patients and sleep analyst) prospective randomized controlled trial to be conducted at Faculty of Dentistry, University of Malaya.

Eligible and consented patients will be randomized into three groups using block randomization with allocation concealment. Patients in Group 1 and 2 will receive MAA set at 25%, 50% of maximum mandibular advancement respectively.

A general medical history will be recorded. Demographic data will be obtained from patients. Baseline measurements will be recorded as T0.

Alginate impressions of the upper and lower dental arches will be taken. Respective mandibular advancement record i.e. at 25% and 50% as assigned by block randomization will be registered using George Gauge. Monobloc type of MAA will then be custom-made for each patient.

Upon issue of MAA, patients will be given detailed instructions for the insertion, removal, storage, and maintenance of MAA. Patients will be advised to wear the MAA every night during sleep. Each patient will be reviewed one week after issue to assess for any problems encountered, adjust the MAA for comfort, and reinforce wear for compliance. Subsequent follow up will be scheduled at every 4-6 weeks. 6 months later, outcome measurements will be recorded as T1.

Baseline and outcome measurements at T0 and T1:

Baseline measurements will be performed prior to intervention (T0) and outcome measurements will be performed 6 months after issue of MAA (T1). Apnea-hypopnea index, minimum oxygen saturation, blood pressure, Epworth Sleepiness Scale(ESS), Calgary Sleep Apnea Quality of Life Index(SAQLI) and dental changes will be measured for both baseline and outcome records. Compliance to MAA and secondary effects caused by MAA will be assessed at T1.

Apnea-Hypopnea Index (AHI), minimum oxygen saturation (Min SaO2) and blood pressure:

AHI and MinSaO2 will be obtained from an overnight polysomnography (PSG) in the sleep laboratory, University of Malaya Medical Center (UMMC). Patient will be instructed to wear the MAA during PSG at T1.

Epworth Sleepiness Scale (ESS):

Daytime sleepiness is to be assessed using ESS. The Malay, Tamil, Mandarin, or English version of the ESS, wherever applicable will be completed by patients.

Calgary Sleep Apnea Quality of Life (SAQLI):

Patient will be interviewed for quality of life assessment using Malay or English version of SAQLI, wherever appropriate.

Compliance to MAA:

Compliance to MAA will be assessed using self-administered diary. Upon issue of MAA, each patient will be given a customized diary to record the frequency of MAA wear daily. The diary will be collected at every review at 4-6 weeks for analysis by calculating the percentage of night per week of wearing the MAA.

Secondary Changes after wearing MAA:

Secondary effect will be evaluated in a structured interview at every review at 4-6 weeks. Temporomandibular joint will be assessed using Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).

Dental Changes after wearing MAA:

Dental changes will be measured with digital caliper and analysed using manual model analysis. The impressions for study models will be taken at T0 and T1.

Blinding:

A single clinician will treat all the patients and one dental technician will make all the MAA. The patient will be blinded to the amount of mandibular advancement. Sleep technician who carries out PSG will also be blinded. Clinician, however, is unable to be blinded due to the need to prescribe the MAA according to the randomization. All the data collected will be coded prior to blinded data analysis.

Proposed Data analysis:

All analyses are to be conducted using SPSS version 25.0. Shapiro-Wilk normality test will be used to evaluate for skewness. Parametric test will be used if the result is assumed normal but if not, non-parametric test will be used instead. Proposed parametric test are paired-sample t tests to test the null hypothesis of no differences AHI, MinSaO2, blood pressure, ESS, SAQLI, compliance and secondary effects, dental changes and demographic baselines between two groups. For the effect of different protrusion amounts and the difference in baseline body mass index(BMI) for both groups, independent T-test will be used instead.

ELIGIBILITY:
Inclusion Criteria:

1. Mild and moderate OSA patients who are keen on MAA
2. Severe OSA who had refuse CPAP
3. Aged 18 years and older
4. Without any form of prior treatment
5. Absence of any structural obstruction examined by otolaryngologist
6. Sufficient set of teeth to hold the appliance

Exclusion Criteria:

1. Presence of periodontal disease
2. Exaggerated gag reflex and temporomandibular joint disorder
3. Significant co-morbidity that could endanger the patient's health
4. Any psychiatric or neurological diseases previously known that could impair the compliance
5. Any medication intake that can influence sleep
6. Co-existing sleep disorders other than OSA for instance insomnia, central sleep apnea and etc
7. Pregnant candidates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea-hypopnea index (AHI) | 6 months
  Apnea Hypopnea Index (AHI) is one of the parameters obtained from polysomnography(PSG) to determine the severity of obstructive sleep apnoea.
  The AHI is the number of apneas or hypopneas recorded during the study per hour of sleep. It is generally expressed as the number of events per hour. Based on the AHI, the severity of OSA is classified as follows:
  None/Minimal: AHI < 5 per hour; Mild: AHI ≥ 5, but < 15 per hour; Moderate: AHI ≥ 15, but < 30 per hour and Severe: AHI ≥ 30 per hour.
  For comparison with other studies, we will also calculate the percentage of patients achieving: (1) reduction in AHI ≥50%; (2) AHI <10; and (3) AHI <5, together with the success criteria defining complete response(CR) as resolution of symptoms and outcome AHI <5, and partial response(PR) as improvement of symptoms and reduction in AHI ≥50% but outcome AHI ≥5. Failure(F) was defined as a reduction in AHI <50% and ⁄ or ongoing symptoms.

SECONDARY OUTCOMES:
Change in Blood Pressure | 6 months
  Compare both systolic and diastolic blood pressure level in pre-treatment and post-treatment
Change in Epworth Sleepiness Scale (ESS) | 6 months
  The ESS is a self-administered questionnaire that evaluates subjective daytime sleepiness. It is usually used as one of the a screening test before sending patients for further evaluation. There are a total of 8 questions. The score ranges from 0 to 24 and is usually raised in sleep apnoea patients, indicating an increased chance to fall asleep. Each question is scored 0 to 3: the total score can vary from 0(no sleepiness) to 24(severe somnolence). A reduction in score would indicate patient has improve condition of alertness.
Change in minimum oxygen saturation (MinSaO2) | 6 months
  Reductions in blood oxygen levels (desaturation) are recorded during polysomnography(PSG).
  At sea level, a normal blood oxygen level (saturation) is usually 96 - 97%. Although there are no generally accepted classifications for severity of oxygen desaturation, reductions to not less than 90% usually are considered mild. Dips into the 80 - 89% range can be considered moderate, and those below 80% are severe.
Change in Quality of Life: Calgary Sleep Apnea Quality of Life Index (SAQLI) | 6 months
  Each of the four SAQLI domains of normal daily routine, social interactions, emotional functioning, and symptoms were similar across strata of disease severity and sex.
  The SAQLI uses a 7-point Likert scale ranging from 1 (maximal impairment) to 7 (no impairment). Domain scores are averaged by dividing by the number of questions answered, and the total score is averaged over the four domains so that all scores maintain a total range of 1 to 7. Unlike other quality of life questionnaires, the SAQLI includes a fifth domain, to capture some of the adverse consequences of currently available therapies for sleep apnoea. This fifth domain, comprising treatment-related symptoms, is used after an intervention, and is subtracted from the other four domains in determining the total SAQLI score.
  The higher the score, the better is the quality of life.
Compliance of wearing the mandibular advancement appliance(MAA) | 6 months
  Compliance will be assessed through compliance diary (percent of nights per week of wearing). Reasons for non-compliance and secondary effects will be evaluated in a structured interview. The stated reasons that lead to non-compliance was investigated.
Secondary effects of wearing mandibular advancement appliance(MAA) | 6 months
  Reasons for non-compliance can be a contributor to secondary effects. The secondary effects caused by mandibular advancement appliance that affects the compliance can be obtained in a structured interview.
  The secondary effect can be excessive salivation, dry mouth, gum irritation, aching of teeth for at least an hour, transient/temporary changes in bite after wake up from sleep, difficulty in chewing in the morning, difficulty in chewing with your back teeth that persist most of the day, appliance frequently dislodge during sleep, difficult to breath through the appliance, pain/aching in jaw joint or jaw muscles and/ or others as suggested by the subjects.
Dental changes after wearing mandibular advancement appliance(MAA)-overjet, overbite, intercanine width, intermolar width and arch length | 6 months
  Dental changes were measured using digital caliper on study models. The electric digital caliper used has an accuracy of 0.01 mm by comparing the study models in overjet, overbite, intercanine width, intermolar width and arch length. Overjet (OJ) is defined as the distance between the upper and lower incisors in the horizontal plane. Overbite (OB) is defined as the vertical overlap of the anterior teeth. Intercanine arch width is the distance between cusp tip points of the right and left canines. Intermolar width is the distance between the mesiobuccal cusp tip points of the first permanent molars. Arch Length is defined as the distance from the line perpendicular to the mesiobuccal cusp tips of the first permanent molars to the midpoint between the mesioincisal points of the central incisors.
Dental changes after wearing mandibular advancement appliance(MAA)-Little's irregularity Index | 6 months
  Dental changes were measured using digital caliper on study models. The electric digital caliper used has an accuracy of 0.01 mm. Little's Irregularity Index is an index used to measure the crowding of mandibular anterior arch. As the crowding increases, the score will increase. The number correspond to the distance in mm of the sum of horizontal displacements of the anatomical contact points of the mandibular anterior teeth. The scale of the index is as listed below.
  0 - Perfect alignment; 1-3 - Minimal irregularity; 4-6 - Moderate irregularity; 7-9 - Severe irregularity and 10 - Very severe irregularity

CONTACTS AND LOCATIONS:
Overall Officials: Lau May Nak, Study Director — University of Malaya
Locations (1):
- Faculty of Dentistry, University of Malaya, Petaling Jaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No